CLINICAL TRIAL: NCT03103919
Title: A Multicenter, Open-Label, Two-Arm Study to Evaluate the Impact of Using Wearable Devices in Addition to Standard Clinical Practice on Parkinson´s Subject Symptoms Management
Brief Title: Study to Evaluate the Impact of Using Wearable Devices in Addition to Standard Clinical Practice on Parkinson´s Subject Symptoms Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PD0049
Record Dates: First submitted 2017-03-30; First posted 2017-04-06 (Actual); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Parkinson´s Disease
Keywords: Parkinson´s Disease; Kinesia-360™; Kinesia-ONE™; Biosensor
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Rotigotine + Standard Care (Active Comparator): Subjects will use the Kinesia-ONE™ wearable device in-clinic at Visit 1 and Visit 2 for recording of specific motor symptoms. The optimal dose of Neupro for any given subject will be determined by standard clinical practice.
  Interventions: Device: Kinesia-ONE™; Drug: Rotigotine
- Rotigotine + Standard Care + Kinesia-360™ wearable device (Experimental): Subjects will use the Kinesia-ONE™ wearable device in-clinic at Visit 1 and Visit 2 for recording of specific motor symptoms, and additionally subjects will use the Kinesia-360™ wearable device at home while awake for continuous measurement of motor symptoms. The Investigator will use these symptom data to provide feedback to subjects on their motor symptoms and to supplement standard of care to titrate the optimal dose of Neupro for any given subject.
  Interventions: Device: Kinesia-ONE™; Device: Kinesia-360™; Drug: Rotigotine

INTERVENTIONS:
Device: Kinesia-ONE™ — Kinesia-ONE™ wearable sensor uses a subject-worn finger sensor and iPad mini application (APP) to objectively measure specific motor tasks related to Parkinson's disease symptoms such as tremor, bradykinesia (slowed movements), and dyskinesia (involuntary movements) in the Investigator's office. Subjects should wear the Kinesia-ONE™ device on the most affected side.
Device: Kinesia-360™ — Kinesia-360™ wearable sensor includes a wrist and ankle device, along with a cell phone, which is also APP-based, and is designed for continuous day time monitoring of Parkinson's disease symptoms. Subjects will wear Kinesia-360™ while they go about their daily lives, and symptom severity is continually captured to enable objective assessment of Parkinson's disease symptoms. Subjects should wear the Kinesia-360™ device bands on the most affected side.
  Arms: Rotigotine + Standard Care + Kinesia-360™ wearable device
Drug: Rotigotine — All subjects will start Neupro treatment at a dose of either rotigotine 2 mg/24 h or 4 mg/24 h (according to the disease stage of the subject) which will then be adjusted based on symptom assessment either via standard care alone or via a combination of standard care and evaluation of the recordings made available by the Kinesia wearable technologies.
  Other Names: Neupro

SUMMARY:
Evaluate the benefits of Kinesia-360™ wearable technology in addition to standard clinical practice on improving Parkinson´s disease motor symptoms, Neupro dosing regimen and adherence to Neupro compared with only standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subject is newly prescribed Neupro and is expected to commence Neupro treatment. Historical Neupro treatment is permitted
* Informed Consent form (ICF) is signed and dated by the subject, before any study-related procedures
* Subject is considered reliable and capable of adhering to the protocol, visit schedule, completion of the diary, and using Kinesia devices according to the judgment of the Investigator
* Male or female subject, >=18 years of age at the time of the Screening Visit
* Subject has Parkinson's disease, defined by the cardinal sign, bradykinesia, plus the presence of at least 1 of the following: tremor at rest, rigidity or impairment of postural reflexes, and without any other known or suspected cause of Secondary Parkinsonism
* Subject experiences motor symptoms associated with Parkinson's disease that are not sufficiently controlled by current therapy. The average of the triplicate resting tremor scores and triplicate finger tapping scores from Kinesia-ONE™ (6 scores in total) must be >1.0

Exclusion Criteria:

* Subject is currently participating in any study with an investigational medicinal product or investigational device
* Subject has any medical, neurological or psychiatric condition which, in the opinion of the Investigator, could jeopardize or would compromise the subject's ability to participate in this study
* Subject with Deep Brain Stimulation (DBS) device implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (8):
- United States (8):
  - Pd0049 105, Fountain Valley, California
  - Pd0049 102, Boca Raton, Florida
  - Pd0049 108, Winfield, Illinois
  - Pd0049 103, Kansas City, Kansas
  - Pd0049 106, Commack, New York
  - Pd0049 104, Tulsa, Oklahoma
  - Pd0049 107, Greenville, South Carolina
  - Pd0049 109, Houston, Texas

REFERENCES:
- See also: Product Information — https://www.neupro.com/neupro-prescribing-information.pdf?v=1489766618
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in March 2017 and concluded in January 2018.
Pre-assignment Details: Participant Flow refers to the Safety Set (SS), which consists of all subjects who received at least 1 dose of Neupro. One subject who received Neupro after screen failing was not considered as treated within the study and, therefore, not included in the SS.
Groups:
- Rotigotine + Standard Care: Subjects used the Kinesia-ONE™ wearable device in-clinic at Visit 1 and Visit 2 for recording of specific motor symptoms. The optimal dose of Neupro for any given subject was determined by standard clinical practice.
- Rotigotine + Standard Care + Kinesia-360™ Wearable Device: Subjects used the Kinesia-ONE™ wearable device in-clinic at Visit 1 and Visit 2 for recording of specific motor symptoms, and additionally subjects used the Kinesia-360™ wearable device at home while awake for continuous measurement of motor symptoms. The Investigator used these symptom data to provide feedback to subjects on their motor symptoms and to supplement standard of care to titrate the optimal dose of Neupro for any given subject.
Period: Overall Study
Arm/Group | Rotigotine + Standard Care | Rotigotine + Standard Care + Kinesia-360™ Wearable Device
Started | 20 | 19
Completed | 18 | 17
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Population: Participant Flow refers to the Safety Set (SS), which consists of all subjects who received at least 1 dose of Neupro. One subject who received Neupro after screen failing was not considered as treated within the study and, therefore, not included in the SS.
Arm/Group | Rotigotine + Standard Care | Rotigotine + Standard Care + Kinesia-360™ Wearable Device | Total Title
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.76 (7.16) | 67.62 (9.77) | 68.72 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 8 | 9 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 2
  White | 17 | 19 | 36
  Other/mixed | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Visit 2 in Unified Parkinson's Disease Rating Scale (UPDRS) Part III Motor Score
Description: UPDRS Part III has 27 items assessing motor skills including facial expression and speech, tremors, rigidity, posture, gait, and bradykinesia. Each of the 27 items in the UPDRS part III is measured on a scale of 0 to 4, where 0 is normal and 4 represents severe abnormalities. The motor score ranges from 0 to 108, where the maximum score indicates the worse condition. A negative value in change in Unified Parkinson's Disease Rating Scale indicates improvement, whereas a positive value indicates worsening of disease.
Time Frame: Baseline (Visit 1/Week 1) to Visit 2 (Week 12/ 3 months after start of treatment with Neupro)
Population: The Full Analysis Set (FAS) included all subjects who had at least 1 valid Baseline and at least 1 valid post-Baseline efficacy measurement.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Groups:
- Rotigotine + Standard Care FAS: Subjects used the Kinesia-ONE™ wearable device in-clinic at Visit 1 and Visit 2 for recording of specific motor symptoms. The optimal dose of Neupro for any given subject was determined by standard clinical practice.
- Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS: Subjects used the Kinesia-ONE™ wearable device in-clinic at Visit 1 and Visit 2 for recording of specific motor symptoms, and additionally subjects used the Kinesia-360™ wearable device at home while awake for continuous measurement of motor symptoms. The Investigator used these symptom data to provide feedback to subjects on their motor symptoms and to supplement standard of care to titrate the optimal dose of Neupro for any given subject.
Arm/Group | Rotigotine + Standard Care FAS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS
Number analyzed (Participants) | 20 | 19
Scores on a scale | -1.0 (2.1) | -5.3 (2.0)
Statistical Analysis 1: Comparison: Rotigotine + Standard Care FAS vs Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS; Test type: Superiority; p = 0.134, ANCOVA; The model used an ANCOVA with baseline as a covariate, center as factor, and group as main factor; Mean Difference (Final Values) = -4.31, 95% CI 2-sided [-10.04 to 1.41] — The difference presented is Experimental Group (Rotigotine + Standard Care + Kinesia-360™ wearable device FAS) minus Control Group (Rotigotine + Standard Care FAS)

2. Primary Outcome: Change From Baseline to Visit 2 in Kinesia-ONE™ Variable: Finger Tapping Speed Score
Description: Kinesia-ONE™ measures were averaged from triplicate repeated assessments at a measurement point. Kinesia-ONE scores ranged from 0 to 4 (where 0 is normal and 4 represents severe abnormalities), with negative change from Baseline scores indicating improvement in disease symptoms.
Time Frame: Baseline (Visit 1/Week 1) to Visit 2 (Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | Rotigotine + Standard Care FAS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS
Number analyzed (Participants) | 19 | 18
Scores on scale | -0.394 (0.160) | -0.389 (0.167)
Statistical Analysis 1: Comparison: Rotigotine + Standard Care FAS vs Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS; Test type: Superiority; p = 0.982, ANCOVA; The model used an ANCOVA with baseline as a covariate, center as factor, and group as main factor; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.44 to 0.45] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Change From Baseline to Visit 2 in Kinesia-ONE™ Variable: Rest Tremor Score
Description: as for outcome 2
Time Frame: Baseline (Visit 1/Week 1) to Visit 2 (Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Rotigotine + Standard Care FAS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS
Number analyzed (Participants) | 19 | 18
Scores on a scale | -0.495 (0.231) | -0.674 (0.238)
Statistical Analysis 1: Comparison: Rotigotine + Standard Care FAS vs Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS; Test type: Superiority; p = 0.566, ANCOVA; The model used an ANCOVA with baseline as a covariate, center as factor, and group as main factor; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.81 to 0.45] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Change From Baseline to Visit 2 in Kinesia-ONE™ Variable: Averaged Finger Tapping Speed and Resting Tremor Scores
Description: Kinesia-ONE™ measures were averaged from triplicate repeated assessments at a measurement point. The finger tapping speed scores and resting tremor scores were averaged and provided as one score ranging from 0 to 4 (where 0 is normal and 4 represents severe abnormalities), with negative change from Baseline scores indicating improvement in disease symptoms.
Time Frame: Baseline (Visit 1/Week 1) to Visit 2 (Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Rotigotine + Standard Care FAS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS
Number analyzed (Participants) | 19 | 18
Scores on a scale | -0.450 (0.156) | -0.525 (0.156)
Statistical Analysis 1: Comparison: Rotigotine + Standard Care FAS vs Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS; Test type: Superiority; p = 0.720, ANCOVA; The model used an ANCOVA with baseline as a covariate, center as factor, and group as main factor; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.50 to 0.35] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Change From Baseline to Visit 2 in Kinesia-ONE™ Variable: Postural Tremor Score
Description: as for outcome 2
Time Frame: Baseline (Visit 1/Week 1) to Visit 2 (Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Rotigotine + Standard Care FAS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS
Number analyzed (Participants) | 19 | 18
Scores on a scale | -0.489 (0.141) | -0.342 (0.143)
Statistical Analysis 1: Comparison: Rotigotine + Standard Care FAS vs Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS; Test type: Superiority; p = 0.443, ANCOVA; The model used an ANCOVA with baseline as a covariate, center as factor, and group as main factor; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.24 to 0.53] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Change From Baseline to Visit 2 in Kinesia-ONE™ Variable: Finger Tapping Amplitude Score
Description: as for outcome 2
Time Frame: Baseline (Visit 1/Week 1) to Visit 2 (Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Rotigotine + Standard Care FAS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS
Number analyzed (Participants) | 19 | 18
Scores on a scale | 0.083 (0.242) | -0.009 (0.238)
Statistical Analysis 1: Comparison: Rotigotine + Standard Care FAS vs Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS; Test type: Superiority; p = 0.777, ANCOVA; The model used an ANCOVA with baseline as a covariate, center as factor, and group as main factor; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.75 to 0.57] — [estimate comment as in outcome 1, analysis 1]

7. Primary Outcome: Change From Baseline to Visit 2 in Kinesia-ONE™ Variable: Hand Grasp Speed Score
Description: as for outcome 2
Time Frame: Baseline (Visit 1/Week 1) to Visit 2 (Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Rotigotine + Standard Care FAS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS
Number analyzed (Participants) | 19 | 18
Scores on a scale | -0.178 (0.115) | -0.188 (0.117)
Statistical Analysis 1: Comparison: Rotigotine + Standard Care FAS vs Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS; Test type: Superiority; p = 0.947, ANCOVA; The model used an ANCOVA with baseline as a covariate, center as factor, and group as main factor; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.33 to 0.31] — [estimate comment as in outcome 1, analysis 1]

8. Primary Outcome: Change From Baseline to Visit 2 in Kinesia-ONE™ Variable: Hand Grasp Amplitude Score
Description: as for outcome 2
Time Frame: Baseline (Visit 1/Week 1) to Visit 2 (Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Rotigotine + Standard Care FAS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS
Number analyzed (Participants) | 19 | 18
Scores on a scale | 0.119 (0.190) | -0.147 (0.188)
Statistical Analysis 1: Comparison: Rotigotine + Standard Care FAS vs Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS; Test type: Superiority; p = 0.306, ANCOVA; The model used an ANCOVA with baseline as a covariate, center as factor, and group as main factor; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.79 to 0.26] — [estimate comment as in outcome 1, analysis 1]

9. Primary Outcome: Change From Baseline to Visit 2 in Kinesia-ONE™ Variable: Rapid Alternating Movement Speed Score
Description: as for outcome 2
Time Frame: Baseline (Visit 1/Week 1) to Visit 2 (Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Rotigotine + Standard Care FAS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS
Number analyzed (Participants) | 19 | 18
Scores on a scale | -0.202 (0.102) | -0.171 (0.106)
Statistical Analysis 1: Comparison: Rotigotine + Standard Care FAS vs Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS; Test type: Superiority; p = 0.819, ANCOVA; The model used an ANCOVA with baseline as a covariate, center as factor, and group as main factor; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.25 to 0.31] — [estimate comment as in outcome 1, analysis 1]

10. Primary Outcome: Change From Baseline to Visit 2 in Kinesia-ONE™ Variable: Rapid Alternating Amplitude Score
Description: as for outcome 2
Time Frame: Baseline (Visit 1/Week 1) to Visit 2 (Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Rotigotine + Standard Care FAS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS
Number analyzed (Participants) | 19 | 18
Scores on a scale | -0.240 (0.123) | -0.167 (0.122)
Statistical Analysis 1: Comparison: Rotigotine + Standard Care FAS vs Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS; Test type: Superiority; p = 0.663, ANCOVA; The model used an ANCOVA with baseline as a covariate, center as factor, and group as main factor; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.26 to 0.41]

11. Primary Outcome: Change From Baseline to Visit 2 in Kinesia-ONE™ Variable: Dyskinesia Score
Description: as for outcome 2
Time Frame: Baseline (Visit 1/Week 1) to Visit 2 (Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Rotigotine + Standard Care FAS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS
Number analyzed (Participants) | 19 | 18
Scores on a scale | 0.125 (0.108) | -0.074 (0.112)
Statistical Analysis 1: Comparison: Rotigotine + Standard Care FAS vs Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS; Test type: Superiority; p = 0.197, ANCOVA; The model used an ANCOVA with baseline as a covariate, center as factor, and group as main factor; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.51 to 0.11]

12. Primary Outcome: Neupro Dose Per 24h at Visit 2 (Week 12)
Description: Daily dose of study medication taken at respective visit.
Time Frame: Visit 2 (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/24 hr
Arm/Group | Rotigotine + Standard Care FAS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device FAS
Number analyzed (Participants) | 16 | 16
mg/24 hr | 3.9 (1.7) | 4.8 (1.8)

13. Primary Outcome: Number of Neupro Dose Changes During the Study
Description: Dose adjustments during study are performed per standard of care.
Time Frame: Visit 1 (Week 1) to Visit 2 (Week 12)
Population: The Safety Set (SS) included all subjects who received at least 1 dose of Neupro.
Measure: Mean (Standard Deviation); unit: dose changes
Groups:
- Rotigotine + Standard Care SS: Subjects used the Kinesia-ONE™ wearable device in-clinic at Visit 1 and Visit 2 for recording of specific motor symptoms. The optimal dose of Neupro for any given subject was determined by standard clinical practice.
- Rotigotine + Standard Care + Kinesia-360™ Wearable Device SS: Subjects used the Kinesia-ONE™ wearable device in-clinic at Visit 1 and Visit 2 for recording of specific motor symptoms, and additionally subjects used the Kinesia-360™ wearable device at home while awake for continuous measurement of motor symptoms. The Investigator used these symptom data to provide feedback to subjects on their motor symptoms and to supplement standard of care to titrate the optimal dose of Neupro for any given subject.
Arm/Group | Rotigotine + Standard Care SS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device SS
Number analyzed (Participants) | 20 | 19
dose changes | 1.8 (1.2) | 2.8 (1.7)

14. Primary Outcome: Number of Subjects Who Discontinued the Treatment With Neupro During the Course of the Study
Description: Number of subjects who discontinued Neupro Treatment were recorded.
Time Frame: Visit 1 (Week 1) to Visit 2 (Week 12)
Population: The Safety Set (SS) included all subjects who received at least 1 dose of Neupro.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotigotine + Standard Care SS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device SS
Number analyzed (Participants) | 20 | 19
Participants | 5 | 5
Statistical Analysis 1: Comparison: Rotigotine + Standard Care SS vs Rotigotine + Standard Care + Kinesia-360™ Wearable Device SS; Test type: Superiority; p = 0.876, Regression, Logistic — P-values for the comparison of treatment groups have been calculated using logistic regression with factors for treatment and center; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.23 to 5.66] — Odds ratio was calculated as Control Group/Experimental Group (Rotigotine + Standard Care SS / Rotigotine + Standard Care + Kinesia-360™ wearable device SS) calculated using logistic regression with factors for treatment and center

15. Secondary Outcome: Number of Subjects With Any Adverse Events During the Course of the Study
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: Visit 1 (Week 1) to Visit 2 (Week 12)
Population: The Safety Set (SS) included all subjects who received at least 1 dose of Neupro.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotigotine + Standard Care SS | Rotigotine + Standard Care + Kinesia-360™ Wearable Device SS
Number analyzed (Participants) | 20 | 19
Participants | 9 | 11

ADVERSE EVENTS:
Time Frame: From Visit 1 (Day 1) to Visit 2 (Week 12)
Arm/Group | Rotigotine + Standard Care | Rotigotine + Standard Care + Kinesia-360™ Wearable Device
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/19
Other Adverse Events (participants affected / at risk) | 9/20 | 10/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine + Standard Care (N=20) | Rotigotine + Standard Care + Kinesia-360™ Wearable Device (N=19)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine + Standard Care (N=20) | Rotigotine + Standard Care + Kinesia-360™ Wearable Device (N=19)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3)
Asthenia (General disorders) | 0 (0) | 2 (2)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 4 (5)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Binge eating (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/19/NCT03103919/SAP_000.pdf
  • Study Protocol (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT03103919/Prot_001.pdf